CLINICAL TRIAL: NCT01753037
Title: Effects of Oral Androgen Administration on Hyperglycemia-Induced Inflammation in Lean Reproductive-Age Women
Brief Title: Effects of Androgen Administration on Inflammation in Normal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Frank Gonzalez, Study Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Mayo-06-004680
Record Dates: First submitted 2012-12-15; First posted 2012-12-20 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2012-12

CONDITIONS: Hyperandrogenism
Keywords: Hyperandrogenism; Inflammation; Insulin sensitivity; Body composition
MeSH Terms: conditions — Hyperandrogenism; Inflammation; Insulin Resistance | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHEA Group (Active Comparator): Oral administration of a capsule containing 130 mg of dehydroepiandrosterone (DHEA) for 5 days.
  Interventions: Dietary Supplement: Dehydroepiandrosterone (DHEA)
- Placebo Group (Placebo Comparator): Oral administration of an identical capsule containing placebo for 5 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dehydroepiandrosterone (DHEA) — DHEA 130 mg administered orally for 5 days.
  Arms: DHEA Group
Other: Placebo — Placebo contained in a capsule that is identical in appearance to the one used to package DHEA for 5 days.
  Arms: Placebo Group

SUMMARY:
The hypothesis of this study is that DHEA administration to increase male hormone in healthy normal-weight young women to levels present in women with Polycystic Ovary Syndrome will cause an inflammatory response in white blood cells in the fasting state, and in response to glucose ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Acceptable health based on interview, medical history, physical examination and lab tests
* Ability to comply with requirements of the study
* Ability and willingness to provide signed, witnessed informed consent
* Between the ages of 18-40 years
* Body mass index between 18 and 25
* Normal regular monthly periods
* No clinical evidence of androgen excess
* No evidence of polycystic ovaries on ultrasound

Exclusion Criteria:

* Diabetes mellitus
* Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious and malignant disease
* High blood pressure
* Current or recent (within 30 days prior to study entry) use of any drugs known or suspected to affect reproductive function including oral contraceptives, metformin, gonadotropin releasing hormone agonists, or anti-androgens (spironolactone, flutamide, etc.)
* Use of medications that have an adverse drug interaction with DHEA therapy including antipsychotics, phenothiazines, lithium, selective serotonin reuptake inhibitors, triazolam, estrogen or testosterone formulations
* Known hypersensitivity to DHEA
* Two first-degree relatives with breast cancer or ovarian cancer
* Documented or suspected history of recent (within 1 year) illicit drug abuse or alcoholism
* Tobacco smoking
* Ingestion of any investigational drugs within 4 weeks prior to study onset
* Pregnancy or lactation (less than or equal to 6 weeks postpartum)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Nuclear factor kappa B (NFkappaB) activation | 0 and 2 hours after glucose ingestion
  White blood cell NFkappaB activation will be assessed in response to glucose ingestion before and after 5 days of DHEA or placebo administration.

SECONDARY OUTCOMES:
Insulin sensitivity | 0 and 5 days after DHEA or placebo
  Insulin sensitivity derived from an oral glucose tolerance test (OGTT) will be assessed before and after 5 days of DHEA or placebo administration.

CONTACTS AND LOCATIONS:
Overall Officials: Frank González, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States